CLINICAL TRIAL: NCT04685499
Title: Phase 2 Study of OBP-301 (Telomelysin ™) in Combination With Pembrolizumab and Stereotactic Body Irradiation in Patients With Head and Neck Squamous Cell Carcinoma With Inoperable, Recurrent or Progressive Disease
Brief Title: Phase 2 Study of OBP-301 (Telomelysin™) in Combination With Pembrolizumab and SBRT in Patients With HNSCC With Inoperable, Recurrent or Progressive Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated due to low participant enrollment.
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Oncolys BioPharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-12021148
Record Dates: First submitted 2020-12-22; First posted 2020-12-28 (Actual); Results first posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2022-12

CONDITIONS: Head and Neck Squamous Cell Carcinoma With Inoperable Recurrent or Progressive Disease
Keywords: Head and Neck; Recurrent; Cure; Unresectable; Immunotherapy; Oncolytic Virus; SBRT; Intratumoral injection
MeSH Terms: conditions — Disease Progression; Recurrence | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Telomelysin (OBP-301) (Experimental): All patients will receive intratumoral injection(s) with OBP-301. If tolerated and no progression is observed, up to twelve injections may be given in each patient.
  Interventions: Drug: OBP-301; Drug: Pembrolizumab

INTERVENTIONS:
Drug: OBP-301 — Telomerase-specific Type 5 Adenovirus. OBP-301 OBP 301 will be injected intratumorally into tumor lesions.
  Other Names: Telomelysin
Drug: Pembrolizumab — Standard dose pembrolizumab 200 mg IV every 3 weeks for up to one year

SUMMARY:
The purpose of this study is to test the effects, of the research study drug Telomelysin (OBP-301) in combination with pembrolizumab in subjects with inoperable, recurrent, or progressive squamous cell carcinoma of the head and neck. Telomelysin is an investigational treatment, while pembrolizumab and SBRT are approved standard treatments. The combination of these three treatments is also considered investigational.

DETAILED DESCRIPTION:
This is a phase II open label single arm study of OBP-301 in combination with pembrolizumab and SBRT in advanced HNSCC which is either recurrent and inoperable, or progressing after prior radiation with curative-intent for advanced disease (adjuvant or definitive with or without chemotherapy or cetuximab).

The efficacy of pembrolizumab monotherapy is modest in second or third line of treatment of advanced head and neck cancer (~response rate 16-22%). SBRT reirradiation in patients that received prior surgery and chemoradiation for advanced disease is associated with a response rate (RR) of approximately 60% and approximately 50% 1-year survival. Recently, the results of the Keynote-048 study were published. The projected 1-year survival in the immunotherapy arms with pembrolizumab alone or pembrolizumab and chemotherapy was approximately 57%. So, at present, the benchmark RR for patients with head and neck squamous cell carcinoma with inoperable, recurrent or progressive disease treated with SBRT is approximately 60% and the 1 year survival for patients with head and neck squamous cell carcinoma (HNSCC) with inoperable, recurrent or progressive disease using the most effective contemporary treatments including immunotherapy is approximately 50-57%. Trying to improve the results of the current standard of care, this study will examine the effects of oncolytic virus, OBP-301, administered in addition to pembrolizumab and SBRT in this patient population. The goal of using this triple therapeutic combination is to enhance the chances of cure of the patients.

A total of 36 patients will be enrolled into a two-stage parallel cohort design: In the first stage, 12 patients will be enrolled.

All patients will receive intratumoral injection(s) with OBP-301. If tolerated and no progression is observed, up to twelve injections may be given in each patient.

If the targeted injected lesion(s) disappear, another lesion can be injected at the Investigator's discretion.

A minimum additional 3 doses of concurrent OBP-301 and pembrolizumab will be given if no toxicity, technical impediment to injection or progression is seen.

A maximum total of up to 9 doses of concurrent OBP-301 and pembrolizumab will be given.

Pembrolizumab alone will be continued after day 183 for a total treatment time up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial.
* Be >18 years of age on the day of signing the informed consent.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Have histologically or cytologically confirmed advanced head and neck squamous cell cancer with cutaneous, subcutaneous or nodal tumors deemed as injectable lesions [see definition below] and have measurable disease for the primary study endpoint of overall response rate by RECIST 1.1 and iRECIST.In addition they must have (A) A single measurable tumor at least 1 cm in size and amenable to intratumoral injection or (B) Multiple measurable tumors that in aggregate have a longest diameter of ≥ 10 mm

Note: Injectable lesion definitions: lesions amenable to percutaneous approach, if technically feasible

* Recurrent and inoperable tumor, progressing after prior radiation with curative-intent for advanced disease (adjuvant or definitive with or without chemotherapy or cetuximab). No prior treatment for local regional recurrence (LRR).
* Tumors may be either HPV+ or HPV-.
* Tumor must be PD-L1 positive, defined as CPS ≥ 1.
* Be willing to provide tissue; newly obtained biopsy specimens or formalin-fixed, paraffin-embedded (FFPE) block specimens.
* Female subjects of childbearing potential have a negative urine or serum pregnancy test within 7 days prior to enrollment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. It is allowed that the test at the same day at 7 days prior to enrollment. And male / female subjects of childbearing potential must agree to use an adequate method of contraception starting with signing the informed consent through 120 days after the last dose of study medication.
* Demonstrated adequate organ function as defined in following criteria. All screening labs should be performed within 14 days of enrollment. Note: Subject must not have taken transfusion, hematopoietic agent; granulocyte-colony stimulating factor (G-CSF) etc., and/or oxygen supplementation within 7 days before the screening labs.

  * Absolute neutrophil count (ANC)>=1,000 /mm3
  * Platelets>=100,000 /mm3
  * Hemoglobin>=9.0 g/dL
  * Serum total bilirubin<=2.0 mg/dL
  * Aspartate aminotransferase (AST) (SGOT) and alanine aminotransferase (ALT) (SGPT) <= 2.5x Upper limit of normal (ULN). For subjects with liver metastases<= 5x ULN.
  * Serum creatinine<= 1.5 mg/dL; or if serum creatinine >1.5 mg/dL, measured or calculated creatinine/clearance>=60 mL/min (Cockcroft-Gault formula).
* Life expectancy of ≥ 6 months from the first OBP-301 treatment.
* Understand the study requirements and the treatment procedures, and is willing to comply with all specified follow- up evaluations, and provides written informed consent before any study-specific tests or procedures are performed.

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy within 2 weeks (chemotherapy, small molecule), or 3 weeks (antibody) of study Day 1.
* Has an active autoimmune disease that has required systemic treatment in past 2 years.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (greater than the equivalent of prednisone 20 mg/day) or any other form of immunosuppressive therapy within 7 days prior to study Day 1. Daily dose of maintenance prednisone 10mg or equivalent is allowable.
* Has known active central nervous system metastases and/or carcinomatous meningitis.
* Has a known additional malignancy that is progressing or requires active treatment, with the exception of stable/low grade tumors that are not expected to influence life-expectancy (e.g. skin SCC, basal cell, differentiated thyroid cancer, prostate cancer on hormonal therapy).
* Has received a live vaccine within 30 days of planned start of study therapy.
* Has a known history of Human Immunodeficiency Virus.
* Has known active Hepatitis B or Hepatitis C.
* Has known history of, or any evidence of active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.
* Previous severe hypersensitivity to another monoclonal antibody.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Prior intolerance related to severe (>=grade 3) irAE to a prior anti-immune checkpoint inhibitor agent leading to discontinuation of anti-immune checkpoint inhibitor therapy.
* Any disorder or condition, or any medication that would put the patient at risk from bleeding after direct tumor injection.
* Not a candidate for SBRT given for potentially curative intent. All tumors must receive SBRT. For example, patients with locoregional neck recurrence without significant overlap with the previous radiation field, and who do not warrant SBRT for re-irradiation as per the treating radiation oncologist (e.g. out-of-field recurrence), will not be included in the study.
* Received prior immunotherapy with checkpoint inhibitors or other immunotherapy agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Doru Paul, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Telomelysin (OBP-301)
Started | 1
Completed | 0
Not Completed | 1
Not completed — Study Terminated Early | 1

BASELINE CHARACTERISTICS:
Arm/Group | Telomelysin (OBP-301)
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate, as Assessed by Radiographic Imaging
Description: Examination of patients with a partial response or complete response.
Time Frame: 30 months
Population: Data not collected.
Arm/Group | Telomelysin (OBP-301)
Number analyzed (Participants) | 0

2. Primary Outcome: Occurrence of Significant Toxicity, as Measured by Number of Grade 3 and Grade 4 Adverse Events (Combined) Attributable to the Combination of Multiple Intratumoral Injections of OBP-301 With SBRT and Pembrolizumab.
Description: We will measure the rate of grade 3 or 4 adverse events attributed to the combination of multiple intratumoral injections of OBP-301 with SBRT and pembrolizumab.
Time Frame: 30 months
Population: Data not collected
Arm/Group | Telomelysin (OBP-301)
Number analyzed (Participants) | 0

3. Secondary Outcome: Disease Control Rate, as Assessed by Radiographic Imaging
Description: Examination of subjects with stable disease, a partial response, or complete response.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Telomelysin (OBP-301)
Number analyzed (Participants) | 1
Participants
  Complete Response | 1
  Partial Response | 0
  Stable Disease | 0

4. Secondary Outcome: Overall Survival, as Measured by the Rate of Survival in Patients
Description: Defined as the time from registration to death from any cause.
Time Frame: 30 months
Population: Data not collected
Arm/Group | Telomelysin (OBP-301)
Number analyzed (Participants) | 0

5. Secondary Outcome: Progression Free Survival, as Assessed by Radiographic Imaging and Survival.
Description: Defined as the time from registration to cancer progression or death due to any cause
Time Frame: 30 months
Population: Data not collected
Arm/Group | Telomelysin (OBP-301)
Number analyzed (Participants) | 0

6. Secondary Outcome: Duration of Response (DoR), as Measured by Subjects Who Have Responded to Combination Therapy Remain Without Disease Progression
Description: defined as the percentage of patients who have achieved complete response, partial response and stable disease.
Time Frame: 30 months
Population: Data not collected.
Arm/Group | Telomelysin (OBP-301)
Number analyzed (Participants) | 0

7. Secondary Outcome: Immune Related Response Rate (irRR), as Assessed by Radiographic Imaging
Description: Examination of subjects with stable disease, a partial response, or complete response.Immune-related disease progression (irPD) will be confirmed if the increase in tumor burden is ≥ 25% relative to nadir (minimum recorded tumor burden).
Time Frame: 30 months
Population: Data not collected
Arm/Group | Telomelysin (OBP-301)
Number analyzed (Participants) | 0

8. Secondary Outcome: Response in Non-target Lesions, as Assessed by Radiographic Imaging
Description: Examination of patients with a partial response or complete response based on RECIST 1.1 and iRECIST
Time Frame: 30 months
Population: Data not collected
Arm/Group | Telomelysin (OBP-301)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: The patient was followed for AEs for 13 months following initiation of treatment.
Arm/Group | Telomelysin (OBP-301)
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telomelysin (OBP-301) (N=1)
Chills (General disorders) | 1 (2)
Headache (General disorders) | 1 (3)
Lightheadedness (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (2)
Diaphoresis (General disorders) | 1 (1)
Hyperkalemia (Investigations) | 1 (1)
Blister (neck) (Skin and subcutaneous tissue disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Aspartate Aminotransferase Increase (Investigations) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-07): https://cdn.clinicaltrials.gov/large-docs/99/NCT04685499/Prot_SAP_000.pdf